CLINICAL TRIAL: NCT00627575
Title: An Open-label, Two-cohort Study to Assess the Effect of Lamotrigine and Phenytoin on the Pharmacokinetics of Atorvastatin in Healthy Subjects
Brief Title: AED/Statin Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LEP108937
Record Dates: First submitted 2008-02-20; First posted 2008-03-03 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Epilepsy
Keywords: drug interaction; pharmacokinetics; healthy volunteers
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine; Atorvastatin; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine (Active Comparator): Subjects will receive 40 milligram (mg) of Atrovastatin from Days 1-7, from Days 8-56 subjects will receive Lamotrigine and Subjects will receive 300 mg/day of Lamotrigine and 40 mg/day of atorvastatin each morning on Days 57-77.
  Interventions: Drug: lamotrigine; Drug: atorvastatin
- phenytoin (Active Comparator): Subjects will receive 40 mg of Atrovastatin from Days 1-7, from Days 8-28, subjects will receive 4mg/kg/day of phenytoin in the morning and will continue to take 40 mg/day of atorvastatin each morning. Subjects will receive taper dose of phenytoin from Days 29-30.
  Interventions: Drug: atorvastatin; Drug: phenytoin

INTERVENTIONS:
Drug: lamotrigine — Lamotrigine tablets will be available in 25, 50, 100 and 200 mg dose strength.
  Arms: Lamotrigine
Drug: atorvastatin — Atorvastatin will available as 40 mg tablets.
Drug: phenytoin — Phenytoin will available as 100 mg capsules.
  Arms: phenytoin

SUMMARY:
This study will evaluate the amount of the cholesterol-lowering drug atorvastatin available in the bloodstream, when taken together with the anti-seizure drugs lamotrigine or phenytoin.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight >50kg (men) or >45kg (women) and BMI within the range 19-32 kg/m2 inclusive.
* No clinically significant abnormality on clinical examination

Key Exclusion Criteria:

* History or evidence of drug or alcohol abuse or active tobacco use.
* Women of childbearing potential
* Use of prescribed or non-prescribed medications during and within 14 days of starting study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2008-02-04 (Actual); Primary Completion 2008-09-12 (Actual); Study Completion 2008-09-12 (Actual)

PRIMARY OUTCOMES:
Steady-state Cmax and AUC (0-t) of atorvastatin | Pre-dose,0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 20 and 24 hrs post dose.
  Steady-state Cmax and AUC (0-t) of atorvastatin when dosed to steady-state.

SECONDARY OUTCOMES:
To assess the effect of lamotrigine or phenytoin on the pharmacokinetics of 2-OH atorvastatin and 4-OH atorvastatin | Pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 20 and 24 hrs post dose.
  Steady state Tmax, Cmax and AUC of 2-OH atorvastatin and 4-OH atorvastatin in the presence and absence of LTG XR or phenytoin.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bullman J, Nicholls A, Van Landingham K, Fleck R, Vuong A, Miller J, Alexander S, Messenheimer J. Effects of lamotrigine and phenytoin on the pharmacokinetics of atorvastatin in healthy volunteers. Epilepsia. 2011 Jul;52(7):1351-8. doi: 10.1111/j.1528-1167.2011.03118.x. Epub 2011 Jun 2. PMID 21635243
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study LEP108937 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/LEP108937?search=study&search_terms=LEP108937#rs
- Available data/document: Clinical Study Report: LEP108937 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LEP108937 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LEP108937 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LEP108937 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LEP108937 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LEP108937 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LEP108937 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register